CLINICAL TRIAL: NCT02919059
Title: A Randomized, Unicenter, Parallel Study of the Effect of Dapagliflozin on Central Blood Pressure Reduction Compared to Glimepiride in Adult Subjects With Type 2 Diabetes Mellitus and Inadequate Glycemic Control.
Brief Title: Study to Asses the Effect of Dapagliflozin on Central Blood Pressure Reduction.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IInstituto Gallego de Medicina Vascular (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESR-14-10158
Record Dates: First submitted 2016-09-23; First posted 2016-09-29 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin 10 mg (Experimental): Dapagliflozin 10 mg once daily during 24 weeks
  Interventions: Drug: Dapagliflozin 10 mg
- Glimepiride 4 mg (Active Comparator): Glimepiride 4 mg once daily during 24 weeks
  Interventions: Drug: Glimepiride 4 mg

INTERVENTIONS:
Drug: Dapagliflozin 10 mg — Dagliflozin will be administred once daily before the first meal of the day for the duration of the study or until early discontinuation. Subjects will take the first dose of study drug at the study centre on Day 1.
  On the day of study visits when fasting blood samples are collected, subjects will be instructed to refrain from taking the study drug before the clinic visit. The subject will be instructed to take the dose of study drug before the subject´s next meal.
  The study drug must be swallowed whole with liquid and not chewed, divided, dissolved or crushed. If the subject doesn´t take the study drug within 12 hours after the first meal of the day, the dose of the study drug should be skipped for that day and keep on taking the study drug on the following day before the first meal.
  Other Names: Dapagliflozin
  Arms: Dapagliflozin 10 mg
Drug: Glimepiride 4 mg — Glimepiride will be administred once daily before the first meal of the day for the duration of the study or until early discontinuation. Subjects will take the first dose of study drug at the study centre on Day 1.
  On the day of study visits when fasting blood samples are collected, subjects will be instructed to refrain from taking the study drug before the clinic visit. The subject will be instructed to take the dose of study drug before the subject´s next meal.
  The study drug must be swallowed whole with liquid and not chewed, divided, dissolved or crushed. If the subject doesn´t take the study drug within 12 hours after the first meal of the day, the dose of the study drug should be skipped for that day and keep on taking the study drug on the following day before the first meal.
  Other Names: Glimepiride
  Arms: Glimepiride 4 mg

SUMMARY:
This superiority of central pressure versus peripheral measures to predict cardiovascular events has also been reported in general population or in elder people

DETAILED DESCRIPTION:
The prognostic value of central systolic/diastolic pressure, central pulse pressure and AI has been well demonstrated, firstly after CAFÉ study, with 2073 hypertensive subjects followed up 3.4 years. It also evidenced higher prognostic value of central blood pressure compared to peripheral blood pressure. One year later, the STRONG study, showed central pulse pressure to be an independent cardiovascular risk factor as well as higher prognostic value compared to peripheral pulse pressure (Hazard ratio; 1,1510 mmHg Vs 1,10mmHg; X2: 13,4; p < 0,001). Those subjects with higher central blood pressure and central pulse pressure showed higher incidence of cardiovascular events. This superiority of central pressure versus peripheral measures to predict cardiovascular events has also been reported in general population or in elder people.

Finally, it has been also reported that dapagliflozin modestly reduces systolic blood pressure in patients with T2DM who were mostly receiving treatment for hypertension. Despite office blood pressure remains the gold standard method for screening, diagnostic and treatment of hypertension, it has been also well demonstrated that ambulatory blood pressure monitoring (ABPM) better estimates cardiovascular risk and target organ damage than office blood pressure. It still remains unclear the effects on 24 hours blood pressure reduction with SGLT-2 inhibitors.

The effects of SGLT2 inhibitors on central blood pressure reduction have not been documented.

ELIGIBILITY:
Inclusion Criteria:

* T2DM subjects with uncontrolled glycaemia, based on HbA1c levels (10% ≥ HbA1c ≥ 7%) at Visit 1.
* Patients may be treated for >3 months with a stable doses of metformin at optimal doses tolerated.
* Participants will be able to give and sign informed consent form.
* Age > 18 years of either gender.

Exclusion Criteria:

* Patients with two or more different oral antihyperglycemic agents.
* HbA 1c levels > 10%.
* Systolic BP >160 mm Hg and/or diastolic BP > 100 mm Hg before randomization.
* History of diabetic ketoacidosis, T1DM, pancreas or beta-cell transplantation or diabetes secondary to any condition.
* History of one or more severe hypoglycaemic episode within 6 months before screening.
* Myocardial infarction, unstable angina pectoris, congestive heart failure, life threatening arrhythmia, history of cerebrovascular accident within 3 months.
* Clinically relevant renal disease; defines if serum creatinine equal or lager than 1.5 mg/dl or eGFR < 60 ml/min/1.73m2, at screening.
* Liver function abnormal: glutamic-oxalacetic transaminase lager than 2 times of upper limit normal or glutamic-pyruvic transaminase lager than 2 times of upper limit normal
* Existence of any serious systemic disease
* Allergic history to the compounds of study medication
* Can not comply the study protocol or misunderstand the informed consent form
* Women of childbearing potential will be required to use a double-barrier method of birth control throughout study participation. Women who are surgically sterile or documented post-menopausal for at least 2 years are not considered to be of childbearing potential.
* Pregnant or breast-feeding or planning to become pregnant during the study.
* History of alcohol abuse (>350 g/week) within 3 years before screening.
* Concurrent therapy with medications that could be affect glycaemia (e.g. corticosteroids) or disallowed therapy (e.g. digoxin).
* Investigational drug treatment within the past 4 months
* Concomitant psychiatric diseases and/or habit/abuse of psychoactive substances
* Predictable lack of co-operation
* Shifts workers
* Employees of the investigator or study centre.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2016-12-13 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Effect of dapagliflozin relative to glimepiride at 24 weeks of treatment period regarding central systolic blood pressure | 24 weeks
  To assess the effect of dapagliflozin relative to glimepiride at 24 weeks of treatment period in subjects with T2DM, with inadequate glycemic control regarding central systolic blood pressure estimated by applanation tonometry

SECONDARY OUTCOMES:
Effect of dapagliflozin relative to glimepiride at 24 weeks regarding central systolic/diastolic blood pressure | 24 weeks
  To assess the effect of dapagliflozin relative to glimepiride at 24 weeks of treatment period in subjects with T2DM, with inadequate glycemic control regarding central systolic/diastolic blood pressure estimated by applanation tonometry.
Effect of dapagliflozin relative to glimepiride at 24 weeks regarding central pulse pressure | 24 weeks
  To assess the effect of dapagliflozin relative to glimepiride at 24 weeks of treatment period in subjects with T2DM, with inadequate glycemic control regarding central pulse pressure estimated by applanation tonometry.
Effect of dapagliflozin relative to glimepiride at 24 weeks of treatment with inadequate glycemic control regarding 24 hours ambulatory systolic/diastolic blood pressure | 24 weeks
  To assess the effect of dapagliflozin relative to glimepiride at 24 weeks of treatment period in subjects with T2DM, with inadequate glycemic control regarding 24 hours ambulatory systolic/diastolic blood pressure.
Type and number of Adverse events in patienteSafety and tolerability of dapagliflozin relative to glimepiride. | 28 weeks
  Type and number of Adverse events to assess the safety and tolerability of dapagliflozin relative to glimepiride.
Effect of dapagliflozin relative to glimepiride at 24 weeks with inadequate glycemic control regarding augmentation pressure | 24 weeks
  To assess the effect of dapagliflozin relative to glimepiride at 24 weeks of treatment period in subjects with T2DM, with inadequate glycemic control regarding augmentation pressure estimated by applanation tonometry.
Effect of dapagliflozin relative to glimepiride at 24 weeks with inadequate glycemic control regarding augmentation index | 24 weeks
  o assess the effect of dapagliflozin relative to glimepiride at 24 weeks of treatment period in subjects with T2DM, with inadequate glycemic control regarding augmentation index estimated by applanation tonometry.

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Hermida, MD, PhD, Study Director — Hospital Nuestra Señora de la Esperanza
Locations (1):
- Hospital Nuestra Señora de la Esperanza, Santiago de Compostela, Galicia, Spain

IPD SHARING:
Plan to Share IPD: No